CLINICAL TRIAL: NCT02334267
Title: Acid-Base Composition With Use of hemoDialysates: the ABChD Trial
Brief Title: Acid-Base Composition With Use of hemoDialysates
Acronym: ABChD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: ABChD
Record Dates: First submitted 2014-12-11; First posted 2015-01-08 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1: GranuFlo (Active Comparator): Study subjects will be randomized to undergo dialysis treatments using GranuFlo, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using acid dialysate concentrations of NaturaLyte for a second weekly hemodialysis treatment. Intervention: blood and dialysate samples will be obtained at specific time points during the dialysis treatments.
  Interventions: Device: Group 1: GranuFlo
- Group 2: NaturaLyte (Active Comparator): Study subjects will be randomized to undergo dialysis treatments using NaturaLyte, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using acid dialysate concentrations of GranuFlo for a second weekly hemodialysis treatment. Intervention: blood and dialysate samples will be obtained at specific time points during the dialysis treatments.
  Interventions: Device: Group 2: NaturaLyte

INTERVENTIONS:
Device: Group 1: GranuFlo — Study subjects will be randomized to undergo dialysis treatments using GranuFlo, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using NaturaLyte, a commercially available acid dialysate concentration for a second weekly hemodialysis treatment. Intervention: blood and dialysate samples will be obtained at specific time points during the dialysis treatments.
  Other Names: GranuFlo 45X
  Arms: Group 1: GranuFlo
Device: Group 2: NaturaLyte — Study subjects will be randomized to undergo dialysis treatments using NaturaLyte, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using GranuFlo, a commercially available acid dialysate concentration for a second weekly hemodialysis treatment. Intervention: blood and dialysate samples will be obtained at specific time points during the dialysis treatments.
  Other Names: NaturaLyte 45X
  Arms: Group 2: NaturaLyte

SUMMARY:
This study is a prospective, single center, single blind (patient and laboratory), randomized, cross-over, two week investigation of intradialytic acid-base kinetics and physiology associated with use of two commercial acid dialysate concentrates in prevalent hemodialysis patients.

DETAILED DESCRIPTION:
Approximately 10-20 prevalent hemodialysis patients will be recruited. Subjects will randomized to receive one weekly hemodialysis treatment using each of the two acetate acid dialysate buffers of NaturaLyte and GranuFlo, which will be assigned in a random fashion. Acetate and bicarbonate concentrations will be assessed before, at eight time points during, and six time points after the completion of hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible to be entered into this study will meet all of the following criteria:

1. Adult female or male patients; age ≥18 years.
2. End stage renal disease (ESRD) patients treated for >90 days with the modality of maintenance hemodialysis and on a stable dialysis prescription for the prior month.
3. Patients utilizing a hemodialysis vascular access of a functioning arteriovenous fistula (AVF) or graft (AVG) during the prior month. The patient's AVF/AVG must be considered in stable functioning condition and not be expected to require any surgical revision/intervention during participation in the trial.
4. Patients with an average spKt/V of ≥1.2 during 30 days prior to screening as determined by historic monthly laboratory adequacy measurements; for patients with only one available spKt/V an average will not be performed. (Note: spKt/V should not be captured from dialysis machine adequacy measurements.)
5. Screening hemoglobin level of ≥9 g/dL, and investigator considers hemoglobin levels to have been clinically stable for at least 30 days.
6. A sodium bicarbonate basic dialysate prescription that has not had any changes for 30 days prior to randomization, and is anticipated to be unchanged during study participation as determined by the investigator.
7. Unchanged heparin dosing regimen for the past 30 days prior to randomization and anticipated unchanged heparin dosing during participation in this clinical trial.
8. No changes two weeks prior to randomization or anticipated changes throughout the study in any phosphate binders, calcium supplements, anticoagulant therapies that are not used for hemodialysis treatment (e.g. warfarin, dabigatran, apixaban, rivaroxaban and acetylsalicylic acid (ASA)), non-dialysate sodium bicarbonate and/or citrate based concomitant medications.
9. If treated with systemic glucocorticoid/corticosteroid medications, no dose changes in the previous two months before randomization, or anticipated dose changes throughout the study duration; the dosing regimen should be consistent with maintenance therapy (i.e. not for an acute or active uncontrolled disease) as determined by the investigator. (Note: this criteria does not pertain to inhaled and/or topical glucocorticoid/corticosteroid therapies)
10. During the two weeks prior to screening, an average of no more than 3.5 kg in pre-dialysis weight gain. In the event greater than 3.5 kg is noted, the investigator will discuss the specific medical history with the Medical Monitor prior to enrollment.
11. Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

Patients that meet any of the following criteria will be ineligible for this study:

1. Patients unable to provide a signed and dated informed consent for this clinical research study.
2. Pregnant or lactating female patients.
3. Females of reproductive potential who do not agree to use a highly effective method of contraception, as determined by the investigator.
4. Missed a scheduled outpatient dialysis treatment within two weeks prior to screening or anticipated to not attend any prescribed hemodialysis treatments during participation in the study.
5. Screening or historic laboratory values of aspartate aminotransferase (AST), alanine transaminase (ALT), and alkaline phosphatase (ALP) levels ≥ 2 times the upper limit of normal. These blood laboratory tests must have been performed within 30 days prior to screening or prior to randomization.
6. A screening or historic laboratory value of total bilirubin >1.9 mg/dL that was collected within 30 days prior to screening or obtained before randomization.
7. Uncontrolled clinically significant blood pressure as determined by the investigator within 30 days prior to screening.
8. Active or recent bleeding disorder within the past 30 days.
9. Screening or historic platelet count <100,000 platelets per microliter (mcL) that was collected within 30 days prior to screening or before randomization.
10. Chronic supplemental oxygen use within 30 days prior to randomization.
11. Current active and significant chronic obstructive pulmonary disease (COPD) as determined by the investigator.
12. Significant residual renal function as determined by the investigator. If the amount of residual renal function is in doubt, a 24 hour urine will be collected during the clinic admission to confirm the creatinine clearance. Decisions will be made after the results have been obtained as to the inclusion of data for these subjects.
13. Active malignancy or a malignancy within the past five years, with exceptions for basal and squamous cell carcinoma.
14. Active and clinically uncontrolled autoimmune disease as determined by the investigator. Subjects with controlled autoimmune diseases must be considered to be clinically stable in the opinion of the investigator (e.g. subjects with systemic lupus erythematosus (SLE) and no recent flares are not excluded). The investigator will consult with the referring physician if it is necessary to confirm the stability of an autoimmune disease.
15. Diagnosed with human immunodeficiency virus (HIV).
16. Diagnosed with congestive heart failure (CHF) class III or IV as classified by the New York Heart Association (NYHA) (refer to Appendix A) within the past 60 days.
17. Planned or anticipated need for any surgical procedures during participation in the study.
18. Current or recent illicit drug use or alcohol abuse as determined by the investigator.
19. Subjects that have any significant medical condition as determined by the investigator, which make her/him ineligible for the study (e.g. clinically significant vomiting on dialysis which affects acid-base status).
20. Any condition as determined by the investigator that would place the subject at an increased risk, or preclude the subject's full compliance with the study procedures and visits.
21. Treatment with an investigational drug, device or intervention within 30 days prior to and during participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Smith, MD, Principal Investigator — Volunteer Research Group and New Orleans Center for Clinical Research
Locations (1):
- Volunteer Research Group and New Orleans Center for Clinical Research, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith WB, Gibson S, Newman GE, Hendon KS, Askelson M, Zhao J, Hantash J, Flanagan B, Larkin JW, Usvyat LA, Thadhani RI, Maddux FW. The dynamics of the metabolism of acetate and bicarbonate associated with use of hemodialysates in the ABChD trial: a phase IV, prospective, single center, single blind, randomized, cross-over, two week investigation. BMC Nephrol. 2017 Aug 29;18(1):273. doi: 10.1186/s12882-017-0683-6. PMID 28851317

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Week 1 GranuFlo and Week 2 NaturaLyte: Study subjects will be randomized to undergo dialysis treatments using GranuFlo, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using acid dialysate concentrations of NaturaLyte for a second weekly hemodialysis treatment. Intervention: serum and dialysate samples will be obtained at specific timepoints during the dialysis treatments.
  GranuFlow: Study subjects will be randomized to undergo dialysis treatments using GranuFlo, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using NaturaLyte, a commercially available acid dialysate concentration for a second weekly hemodialysis treatment. Intervention: serum and dialysate samples will be obtained at specific timepoints during the dialysis treatments.
- Group 2 Week 1 NaturaLyte and Week 2 GranuFlo: Study subjects will be randomized to undergo dialysis treatments using NaturaLyte, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using acid dialysate concentrations of GranuFlo for a second weekly hemodialysis treatment. Intervention: serum and dialysate samples will be obtained at specific timepoints during the dialysis treatments.
  NaturaLyte: Study subjects will be randomized to undergo dialysis treatments using NaturaLyte, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using GranuFlo, a commercially available acid dialysate concentration for a second weekly hemodialysis treatment. Intervention: serum and dialysate samples will be obtained at specific timepoints during the dialysis treatments.
Period: Overall Study
Arm/Group | Group 1 Week 1 GranuFlo and Week 2 NaturaLyte | Group 2 Week 1 NaturaLyte and Week 2 GranuFlo
Started | 6 | 5
Completed | 5 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1Week 1 GranuFlo and Week 2 NaturaLyte: Study subjects will be randomized to undergo dialysis treatments using GranuFlo, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using acid dialysate concentrations of NaturaLyte for a second weekly hemodialysis treatment. Intervention: serum and dialysate samples will be obtained at specific timepoints during the dialysis treatments.
  GranuFlow: Study subjects will be randomized to undergo dialysis treatments using GranuFlo, a commercially available acid dialysate concentrations for one weekly hemodialysis treatment. This will be followed by dialysis treatments using NaturaLyte, a commercially available acid dialysate concentration for a second weekly hemodialysis treatment. Intervention: serum and dialysate samples will be obtained at specific timepoints during the dialysis treatments.
- Total: Total of all reporting groups
Arm/Group | Group 1Week 1 GranuFlo and Week 2 NaturaLyte | Group 2 Week 1 NaturaLyte and Week 2 GranuFlo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Peridialytic Arterialized Blood Bicarbonate Concentrations
Description: Quantification of Peridialytic Arterialized Blood Bicarbonate Concentrations
Time Frame: Immediately prior to initiation of hemodialysis, and 25, 60, 90, 120, 150, 180, 210, 240 minutes of hemodialysis and 15, 30, 45, 60, 75, and 90 minutes post hemodialysis
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: mEq/l
Groups:
- GranuFlo: The outcome measure was peridialytic arterialized blood bicarbonate concentrations over time in subjects who received a hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate GranuFlo
- NaturaLyte: The outcome measure was peridialytic arterialized blood bicarbonate concentrations over time in subjects who received a hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate NaturaLyte
Arm/Group | GranuFlo | NaturaLyte
Number analyzed (Participants) | 10 | 10
mEq/l
  Pre-dialysis | 25.7 (3.33) | 27.1 (3.28)
  25 min of dialysis | 27.2 (3.16) | 27.4 (3.69)
  60 min of dialysis | 28.9 (3.48) | 28.4 (4.20)
  90 min of dialysis | 29.2 (3.85) | 28.6 (4.14)
  120 min of dialysis | 29.3 (3.89) | 28.3 (3.95)
  150 min of dialysis | 29.2 (3.77) | 28.3 (3.80)
  180 min of dialysis | 29.6 (4.09) | 28.3 (3.71)
  210 min of dialysis | 30.1 (3.90) | 29.1 (3.90)
  240 min of dialysis | 30.2 (4.16) | 28.8 (4.26)
  15 min post-dialysis | 30.8 (4.34) | 29.9 (4.18)
  30 min post-dialysis | 30.9 (4.28) | 29.8 (4.21)
  45 min post-dialysis | 31.2 (3.91) | 29.8 (4.26)
  60 min post-dialysis | 31.4 (3.64) | 30.5 (4.60)
  75 min post-dialysis | 31.6 (4.10) | 29.6 (4.27)
  90 min post-dialysis | 31.2 (4.44) | 29.8 (4.37)
Statistical Analysis 1: Comparison: GranuFlo vs NaturaLyte; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — trend analysis over time

2. Primary Outcome: Peridialytic Venous Blood Bicarbonate Concentrations
Description: Quantification of Peridialytic Venous Blood Bicarbonate Concentrations
Time Frame: 25, 60, 90, 120, 150, 180, 210, 240 minutes of hemodialysis
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: mEq/l
Groups:
- GranuFlo: The outcome measure was peridialytic venous blood bicarbonate concentrations over time in subjects who received a hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate GranuFlo
- NaturaLyte: The outcome measure was peridialytic venous blood bicarbonate concentrations over time in subjects who received a hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate NaturaLyte
Arm/Group | GranuFlo | NaturaLyte
Number analyzed (Participants) | 10 | 10
mEq/l
  25 min of dialysis | 29.4 (3.13) | 30.8 (3.71)
  60 min of dialysis | 30.7 (3.83) | 30.7 (3.89)
  90 min of dialysis | 30.2 (3.36) | 31.2 (3.71)
  120 min of dialysis | 30.7 (3.30) | 30.6 (3.69)
  150 min of dialysis | 30.8 (3.58) | 30.4 (3.84)
  180 min of dialysis | 31.0 (3.83) | 31.3 (3.65)
  210 min of dialysis | 30.3 (3.94) | 31.0 (3.89)
  240 min of dialysis | 30.6 (3.92) | 30.9 (3.96)
Statistical Analysis 1: Comparison: GranuFlo vs NaturaLyte; Test type: Superiority or Other; p = 0.4, Mixed Models Analysis — trend analysis over time

3. Primary Outcome: Peridialytic Arterialized Blood Acetate Concentrations
Description: Quantification of Peridialytic Arterialized Blood Acetate Concentrations
Time Frame: as for outcome 1
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- GranuFlo: The outcome measure was peridialytic arterialized blood acetate concentrations over time in subjects who received a hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate GranuFlo
- NaturaLyte: The outcome measure was peridialytic arterialized blood acetate concentrations over time in subjects who received a hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate NaturaLyte
Arm/Group | GranuFlo | NaturaLyte
Number analyzed (Participants) | 10 | 10
mmol/L
  Pre-dialysis | 0.4 (0.35) | 0.4 (0.32)
  25 min of dialysis | 0.5 (0.29) | 0.4 (0.28)
  60 min of dialysis | 0.3 (0.22) | 0.2 (0.12)
  90 min of dialysis | 0.4 (0.57) | 0.1 (0.12)
  120 min of dialysis | 0.3 (0.18) | 0.1 (0.18)
  150 min of dialysis | 0.2 (0.18) | 0.1 (0.12)
  180 min of dialysis | 0.2 (0.20) | 0.1 (0.11)
  210 min of dialysis | 0.3 (0.21) | 0.2 (0.31)
  240 min of dialysis | 0.4 (0.58) | 0.2 (0.21)
  15 min post-dialysis | 0.0 (0.05) | 0.1 (0.13)
  30 min post-dialysis | 0.1 (0.28) | 0.1 (0.17)
  45 min post-dialysis | 0.2 (0.35) | 0.1 (0.24)
  60 min post-dialysis | 0.6 (1.05) | 0.2 (0.27)
  75 min post-dialysis | 0.4 (0.61) | 0.6 (0.74)
  90 min post-dialysis | 0.4 (0.61) | 0.4 (0.57)
Statistical Analysis 1: Comparison: GranuFlo vs NaturaLyte; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — trend analysis over time

4. Primary Outcome: Peridialytic Venous Blood Acetate Concentrations
Description: Quantification of Peridialytic Venous Blood Acetate Concentrations
Time Frame: 25, 60, 90, 120, 150, 180, 210, 240 minutes of hemodialysis
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- GranuFlo: The outcome measure was peridialytic venous blood acetate concentrations over time in subjects who received a hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate GranuFlo
- NaturaLyte: The outcome measure was peridialytic venous blood acetate concentrations over time in subjects who received a hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate NaturaLyte
Arm/Group | GranuFlo | NaturaLyte
Number analyzed (Participants) | 10 | 10
mmol/L
  25 min of dialysis | 1.7 (0.62) | 1.0 (0.48)
  60 min of dialysis | 1.6 (0.60) | 1.0 (0.52)
  90 min of dialysis | 1.6 (0.81) | 0.9 (0.62)
  120 min of dialysis | 2.0 (0.74) | 1.0 (0.82)
  150 min of dialysis | 1.8 (0.67) | 1.1 (0.65)
  180 min of dialysis | 1.8 (0.70) | 1.1 (0.76)
  210 min of dialysis | 1.9 (0.83) | 1.1 (0.85)
  240 min of dialysis | 1.7 (0.90) | 1.2 (0.84)
Statistical Analysis 1: Comparison: GranuFlo vs NaturaLyte; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — trend analysis over time

ADVERSE EVENTS:
Groups:
- GranuFlo: The safety reporting group included subjects who received one study related hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate GranuFlo.
- NaturaLyte: The safety reporting group included subjects who received one study related hemodialysis treatment with a hemodialysate solution that was made from the acid dialysate concentrate NaturaLyte.
Arm/Group | GranuFlo | NaturaLyte
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GranuFlo (N=10) | NaturaLyte (N=11)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less